CLINICAL TRIAL: NCT01621438
Title: Influence of Total Atherosclerotic Burden Assessed by 3-vessel Fractional Flow Reserve (FFR) on the Clinical Outcomes of the Patients With Multi-vessel Disease
Brief Title: Clinical Implication of 3-vessel Fractional Flow Reserve (FFR)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Samsung Medical Center (Other); Keimyung University Dongsan Medical Center (Other); Inje University (Other); Fu Wai Hospital, Beijing, China (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Guangdong Provincial People's Hospital (Other); Tokyo medical college hospital, Japan (Unknown); Kokura Memorial Hospital (Other); Gifu Heart Center (Other); Aichi Medical University (Other); Wakayama Medical University (Other); Queen Mary Hospital, Hong Kong (Other); United Christian Hospital (Other); National University Heart Centre, Singapore (Other); National Taiwan University Hospital (Other); Nagoya Daini Nesseki Hospital (Other); Ulsan University Hospital (Other); Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Bon-Kwon Koo, Professor, Seoul National University Hospital
Other Study IDs: H-1203-087-402
Record Dates: First submitted 2012-06-07; First posted 2012-06-18 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Multivessel Coronary Artery Disease
Keywords: coronary artery; atherosclerosis; angina pectoris
MeSH Terms: conditions — Atherosclerosis; Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study will evaluate the influence of total atherosclerotic burden assessed by 3-vessel fractional flow reserve (FFR) on the clinical outcomes of the patients with multi-vessel disease. For this purpose, the clinical data of the patients with 3-vessel intermediate coronary artery disease, whose FFR was measured at all 3-vessels due to their own clinical needs, will be analyzed.

DETAILED DESCRIPTION:
Primary Analysis The Primary Analysis will be performed after 2-year follow-up data will be completed.

Pre-specified Subgroup Analysis

The pre-specified subgroup analysis will perform after 1-year follow-up data will be completed according to the following subjects:

* Concordant and discordant results between FFR and angiographic stenosis severity (patients and lesions with pre-PCI FFR will be analyzed.).

  * Association between total atherosclerotic burden and total ischemic burden, coronary CT angiography substudy (after 2-year follow-up will be completed).

    * Validation of total ischemic burden (sum of 3 vessel FFR) with Duke score, measured by treadmill test.

      * Comparison of clinical outcomes of deferred lesions according to pre-PCI FFR levels (Pre-PCI FFR <0.75, 0.75-0.80, and >0.80).

        * Comparison of clinical outcomes of deferred lesions according to iFR and FFR values ⑥ Prognosis of functional complete revascularization versus incomplete revascularization

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age.
* Subject must have stenosis (>30% by visual estimate) in all 3-epicardial coronary arteries.
* FFR should be measured at all 3-vessels at the end of a procedure.

Exclusion Criteria:

* Depressed left ventricular systolic function (ejection fraction < 35%)
* ST-elevation myocardial infarction within 72 hours,
* Prior coronary artery bypass graft surgery
* Creatinine level >= 2.0mg/dL or dependence on dialysis
* Abnormal final myocardial flow (TIMI flow < 3)
* Planned bypass surgery
* Failed FFR measurement
* Failed intended revascularization

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients with 3-vessel intermediate coronary artery disease (visually 30~70% stenosis in coronary angiogram) whose FFR was measured at all 3-vessels due to their own clinical needs.
Sampling Method: Probability Sample
Enrollment: 1136 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-03 (Actual); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
The rate of the composite of major adverse cardiac events (MACE: cardiac death, myocardial infarction, revascularization) at 2 years per 3-vessel FFR | 2 years after FFR measurement

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, MD, Principal Investigator — Cardiovascular Center, Seoul National University Hospital, 101 Daehak-ro, Jongno-gu, Seoul, 110-744, South Korea
Locations (20):
- China (6):
  - Fuwai hospital, Beijing
  - Guandong general hospital, Guandong
  - Queen Mary Hospital, The University of Hong Kong, Hong Kong
  - United Christian Hospital, Hong Kong
  - Nanjing 1st hospital, Nanjing
  - Zhejiang No 2 hospital, Zhejiang
- Japan (6):
  - Gifu heart center, Gifu
  - Kokura memorial hospital, Kitakyushu
  - 2nd Red Cross hospital, Kyoto
  - Aichi Medical university hospital, Nagakute
  - Tokyo medical college hospital, Tokyo
  - Wakayama medical university, Wakayama
- National University Heart center, Singapore, Singapore
- South Korea (6):
  - Keimyung University Dongsan medical center, Daegu
  - Inje university Ilsan Paik hospital, Ilsan
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul, Korea, Seoul
  - Ajou university hospital, Suwon
  - Ulsan university hospital, Ulsan
- National Taiwan University hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Lee JM, Lee SH, Hwang D, Rhee TM, Choi KH, Kim J, Park J, Kim HY, Jung HW, Cho YK, Yoon HJ, Song YB, Hahn JY, Nam CW, Shin ES, Doh JH, Hur SH, Koo BK. Long-Term Clinical Outcomes of Nonhyperemic Pressure Ratios: Resting Full-Cycle Ratio, Diastolic Pressure Ratio, and Instantaneous Wave-Free Ratio. J Am Heart Assoc. 2020 Sep 15;9(18):e016818. doi: 10.1161/JAHA.120.016818. Epub 2020 Sep 11. PMID 32914672
- [Derived] Lee JM, Choi KH, Koo BK, Park J, Kim J, Hwang D, Rhee TM, Kim HY, Jung HW, Kim KJ, Yoshiaki K, Shin ES, Doh JH, Chang HJ, Cho YK, Yoon HJ, Nam CW, Hur SH, Wang J, Chen S, Kuramitsu S, Tanaka N, Matsuo H, Akasaka T. Prognostic Implications of Plaque Characteristics and Stenosis Severity in Patients With Coronary Artery Disease. J Am Coll Cardiol. 2019 May 21;73(19):2413-2424. doi: 10.1016/j.jacc.2019.02.060. PMID 31097161
- [Derived] Kim CH, Koo BK, Lee JM, Shin ES, Park J, Choi KH, Hwang D, Rhee TM, Zhang J, Choi YJ, Lee SY, Choi JH, Doh JH, Nam CW, Wang J, Chen S, Kuramitsu S, Tanaka N, Matsuo H, Akasaka T. Influence of Sex on Relationship Between Total Anatomical and Physiologic Disease Burdens and Their Prognostic Implications in Patients With Coronary Artery Disease. J Am Heart Assoc. 2019 Mar 5;8(5):e011002. doi: 10.1161/JAHA.118.011002. PMID 30813812
- [Derived] Lee JM, Choi KH, Park J, Hwang D, Rhee TM, Kim J, Park J, Kim HY, Jung HW, Cho YK, Yoon HJ, Song YB, Hahn JY, Nam CW, Shin ES, Doh JH, Hur SH, Koo BK. Physiological and Clinical Assessment of Resting Physiological Indexes. Circulation. 2019 Feb 12;139(7):889-900. doi: 10.1161/CIRCULATIONAHA.118.037021. PMID 30586749
- [Derived] Park J, Lee JM, Koo BK, Shin ES, Nam CW, Doh JH, Hwang D, Zhang J, Hu X, Wang J, Ye F, Chen S, Yang J, Chen J, Tanaka N, Yokoi H, Matsuo H, Takashima H, Shiono Y, Akasaka T. Clinical Relevance of Functionally Insignificant Moderate Coronary Artery Stenosis Assessed by 3-Vessel Fractional Flow Reserve Measurement. J Am Heart Assoc. 2018 Feb 15;7(4):e008055. doi: 10.1161/JAHA.117.008055. PMID 29449274
- [Derived] Choi KH, Lee JM, Koo BK, Nam CW, Shin ES, Doh JH, Rhee TM, Hwang D, Park J, Zhang J, Kim KJ, Hu X, Wang J, Ye F, Chen S, Yang J, Chen J, Tanaka N, Yokoi H, Matsuo H, Takashima H, Shiono Y, Akasaka T. Prognostic Implication of Functional Incomplete Revascularization and Residual Functional SYNTAX Score in Patients With Coronary Artery Disease. JACC Cardiovasc Interv. 2018 Feb 12;11(3):237-245. doi: 10.1016/j.jcin.2017.09.009. Epub 2018 Jan 17. PMID 29361444
- [Derived] Kobayashi Y, Lee JM, Fearon WF, Lee JH, Nishi T, Choi DH, Zimmermann FM, Jung JH, Lee HJ, Doh JH, Nam CW, Shin ES, Koo BK. Three-Vessel Assessment of Coronary Microvascular Dysfunction in Patients With Clinical Suspicion of Ischemia: Prospective Observational Study With the Index of Microcirculatory Resistance. Circ Cardiovasc Interv. 2017 Nov;10(11):e005445. doi: 10.1161/CIRCINTERVENTIONS.117.005445. PMID 29146670
- [Derived] Lee JM, Koo BK, Shin ES, Nam CW, Doh JH, Hu X, Ye F, Chen S, Yang J, Chen J, Tanaka N, Yokoi H, Matsuo H, Takashima H, Shiono Y, Hwang D, Park J, Kim KJ, Akasaka T, Wang J. Clinical Outcomes of Deferred Lesions With Angiographically Insignificant Stenosis But Low Fractional Flow Reserve. J Am Heart Assoc. 2017 Aug 22;6(8):e006071. doi: 10.1161/JAHA.117.006071. PMID 28862970
- [Derived] Lee JM, Kim CH, Koo BK, Hwang D, Park J, Zhang J, Tong Y, Jeon KH, Bang JI, Suh M, Paeng JC, Cheon GJ, Na SH, Ahn JM, Park SJ, Kim HS. Integrated Myocardial Perfusion Imaging Diagnostics Improve Detection of Functionally Significant Coronary Artery Stenosis by 13N-ammonia Positron Emission Tomography. Circ Cardiovasc Imaging. 2016 Sep;9(9):e004768. doi: 10.1161/CIRCIMAGING.116.004768. PMID 27609817